CLINICAL TRIAL: NCT00850330
Title: Transversal, Multicentric Study for Early Detection of Drug Interactions in Older Hospitalized Patients Using on Line Software in Córdoba, Argentina
Brief Title: Study for Early Detection of Drug Interactions in Older Hospitalized Patients Using on Line Software
Acronym: SEDDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad Nacional de Córdoba (Other)
Responsible Party: Gabriel Santino Iraci, Catedra de Farmacología. Hospital Nacional de Clínicas. Universidad Nacional de Cordoba
Other Study IDs: Iraci-01
Record Dates: First submitted 2009-02-20; First posted 2009-02-25 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Drug Interactions
Keywords: Drug interactions; Drug interaction software; Older patients; Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized patients: Patients elder than 65 years old hospitalized for any reason.
  Interventions: Other: on line software to detect DI early on

INTERVENTIONS:
Other: on line software to detect DI early on — Patients hospital records will be reviewed on the day of admission to assess all their indication using on line software to early detect drug interactions.
  Other Names: Software are available on:; http://www.medscape.com/druginfo/druginterchecker; http://www.medicamentosrothlin.com.ar/

SUMMARY:
A drug interaction (DI) is the mutual action of two drugs in a way that they can increase their action, even to a toxic level, or reduce it to its minimum.

People elder than 65 years old have theirs biological ability to metabolized and eliminate drugs impaired. Even more, they tend to suffer from many diseases, are treated for many physicians, and receive many drugs for those conditions. If hospitalized older people are prone to receive a greater number of drugs. This scenario is the worst to suffer from adverse drug events and DI, which in turn compromise more the health and even life of hospitalized older people.

Many computerized strategies have been developed to prevent those problems. In this trial the investigators use on line software to early detect DI that could endanger health or life of hospitalized older patients.

DETAILED DESCRIPTION:
A drug interaction (DI) is the mutual action of two drugs in a way that they can increase their action, even to a toxic level, o reduce it to its minimum.

Adverse drug events (ADE) are an important health problem. In the book To Err Is Human: Building a Safer Health System its authors Kohn, Corrigan and Donaldson from the "Committee on Quality of Health Care in America, Institute of Medicine" (U.S.A.) expressed that 2 out of every 100 hospital admissions were due to ADE. That results in an average increase of U$D 4,700 extra for each admission or about to 2.8 million U$D annually for a 700-bed teaching hospital. In this study were only considered direct costs. No indirect costs were taken into account, like days out of work, rehabilitation, deaths, lost of quality of life, etc.

In 2003, in a cohort study done in people of Medicare elder than 65 years old, were detected 50.1 ADE / 1000 persons a year. Of that number of ADE 13.8 were considered preventable. In Switzerland 3.3 % of hospitalisations were considered due to ADE.

Among ADE, DI are a very important part of the problem. In Canada was demonstrated that certain drug associations were responsible of an increase in the number of hospital admissions. They would not have occurred if those prescriptions would have been properly controlled or never done. In Mexico 3.8 % of patients elder than 50 years old received prescriptions of drugs, which should be avoided according to their interaction. In hospital setting DI endanger even more health and people's life. In Spain was demonstrated a prevalence of clinical relevant DI of 3 % in hospitalized patients, and in Switzerland that percentage rose 11 %. This phenomenon increased in later years, in Rotterdam DI compromising lethal risk in patients elder than 70 years old, climb from 1.5 % in 1992 to 2.9 % in 2005. Drug interactions are directly proportional to: the number of administered drugs (> 2 drugs or > 4 ); the age of patients and the number of prescribing physicians.

Older persons, for its detriment in physical condition and the pathologies they suffer from, are prone to suffer DI when being prescribed with drugs or even herbal medicines. In Brazil ambulatory patients elder than 60 years old have 2.5 pathologies diagnosed and consume in average 1.3 to 2.3 drugs. During hospitalisation the number of prescribed drugs reach 9.9 to 13.6 per patient. In a survey done in six European countries the number of drugs consumed for each ambulatory patient was 7. In Argentina according to the Instituto Nacional de Estadísticas y Censos (INDEC) the number of citizens elder than 65 years old was 3,587,620 (9.89% total population). Unfortunately there is no other information about polypharmacy or prevalent pathologies in INDEC or other medical databases or national institutions web sites.

In 1995, it was published an article in JAMA that stated the possibility that 28 % of ADE could be prevented in non-obstetric hospitalized adults. Fifty six percent of those were due to mistakes done during prescription, 34 % during administration, 6 % during transcription of indications and 4 % during dispensation. This astonishing results poses on the need to develop strategies to cut this numbers.

Many lists of drugs with potential to produce ADE were developed to prevent DI and other related drugs damages. Beers criteria (BC) is one example of them. In Amsterdam it was demonstrated an 80 % improvement in drug regimens in patients elder than 81 years old of in whom their therapeutic indications were reviewed and adjusted using BC and the Medication Appropriateness Index after suffering from ADE. In that study, a list of only 10 drug combinations was also used but did not showed the same benefits. In Argentina, the Adminstración Nacional de Medicamentos, Alimentos y Tecnología (ANMAT) publish in its web page a list of 16 risky drugs, considering the disadvantages of their own pharmacological action, but there is no information about its usefulness.

Much software was developed in later years to alert physician about DI. Some of them are even more sensible than the search of DI at the bedside, but this software overestimates the prevalence of serious DI. The usage of computerized alert systems for prescriptions significantly reduced potential ADE, however many physicians tend to override them for different reasons. Finally a Cochrane´s review showed a reduction in hospitalization days and drug toxic effects when using a computerized warning systems for drug dosing.

The growing number of drugs, apart from its not always well-proven benefits, implies risks for health; specially in sick and older people and even more during hospitalizations. Nowadays software to alert physicians about DI or ADE could help to prevent them but its real contribution is still a matter of debate. For this reasons we developed this trial to test the usefulness of on line software to detect DI in hospitalized elder patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization
* 65 years old or more

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patients older than 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Early detect DI in hospitalized elder patients | One year and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel S Iraci, MD, Prof, Principal Investigator — Catedra de Farmacología, Hospital Nacional de Clínicas, Universidad Nacional de Córdoba
Locations (2):
- Argentina (2):
  - Clínica Privada Colombo, Córdoba, Córdoba Province
  - Hospital Nacional de Clínicas, Córdoba, Córdoba Province

REFERENCES:
- [Background] Gurwitz JH, Field TS, Harrold LR, Rothschild J, Debellis K, Seger AC, Cadoret C, Fish LS, Garber L, Kelleher M, Bates DW. Incidence and preventability of adverse drug events among older persons in the ambulatory setting. JAMA. 2003 Mar 5;289(9):1107-16. doi: 10.1001/jama.289.9.1107. PMID 12622580
- [Background] Fattinger K, Roos M, Vergeres P, Holenstein C, Kind B, Masche U, Stocker DN, Braunschweig S, Kullak-Ublick GA, Galeazzi RL, Follath F, Gasser T, Meier PJ. Epidemiology of drug exposure and adverse drug reactions in two swiss departments of internal medicine. Br J Clin Pharmacol. 2000 Feb;49(2):158-67. doi: 10.1046/j.1365-2125.2000.00132.x. PMID 10671911
- [Background] Juurlink DN, Mamdani M, Kopp A, Laupacis A, Redelmeier DA. Drug-drug interactions among elderly patients hospitalized for drug toxicity. JAMA. 2003 Apr 2;289(13):1652-8. doi: 10.1001/jama.289.13.1652. PMID 12672733
- [Background] Doubova Dubova SV, Reyes-Morales H, Torres-Arreola Ldel P, Suarez-Ortega M. Potential drug-drug and drug-disease interactions in prescriptions for ambulatory patients over 50 years of age in family medicine clinics in Mexico City. BMC Health Serv Res. 2007 Sep 19;7:147. doi: 10.1186/1472-6963-7-147. PMID 17880689
- [Background] Peral Aguirregoitia J, Lertxundi Etxebarria U, Martinez Bengoechea MJ, Mora Atorrasagasti O, Franco Lamela E, Gabilondo Zelaia I. [Prospective assessment of drug interactions in hospitalized patients using a computer programme]. Farm Hosp. 2007 Mar-Apr;31(2):93-100. doi: 10.1016/s1130-6343(07)75719-7. Spanish. PMID 17590117
- [Background] Becker ML, Visser LE, van Gelder T, Hofman A, Stricker BH. Increasing exposure to drug-drug interactions between 1992 and 2005 in people aged > or = 55 years. Drugs Aging. 2008;25(2):145-52. doi: 10.2165/00002512-200825020-00006. PMID 18257601
- [Background] Preskorn SH, Silkey B, Shah R, Neff M, Jones TL, Choi J, Golbeck AL. Complexity of medication use in the Veterans Affairs healthcare system: Part I: Outpatient use in relation to age and number of prescribers. J Psychiatr Pract. 2005 Jan;11(1):5-15. doi: 10.1097/00131746-200501000-00002. PMID 15650617
- [Background] Marin MJ, Cecilio LC, Perez AE, Santella F, Silva CB, Goncalves Filho JR, Roceti LC. [Use of medicines by the elderly in a Family Health Program unit in Brazil]. Cad Saude Publica. 2008 Jul;24(7):1545-55. doi: 10.1590/s0102-311x2008000700009. Portuguese. PMID 18670678
- [Background] Medeiros-Souza P, Santos-Neto LL, Kusano LT, Pereira MG. Diagnosis and control of polypharmacy in the elderly. Rev Saude Publica. 2007 Dec;41(6):1049-53. doi: 10.1590/s0034-89102006005000050. Epub 2007 Dec 4. PMID 17992356
- [Background] Bjorkman IK, Fastbom J, Schmidt IK, Bernsten CB; Pharmaceutical Care of the Elderly in Europe Research (PEER) Group. Drug-drug interactions in the elderly. Ann Pharmacother. 2002 Nov;36(11):1675-81. doi: 10.1345/aph.1A484. PMID 12398558
- [Background] Bates DW, Cullen DJ, Laird N, Petersen LA, Small SD, Servi D, Laffel G, Sweitzer BJ, Shea BF, Hallisey R, et al. Incidence of adverse drug events and potential adverse drug events. Implications for prevention. ADE Prevention Study Group. JAMA. 1995 Jul 5;274(1):29-34. PMID 7791255
- [Background] Fick DM, Cooper JW, Wade WE, Waller JL, Maclean JR, Beers MH. Updating the Beers criteria for potentially inappropriate medication use in older adults: results of a US consensus panel of experts. Arch Intern Med. 2003 Dec 8-22;163(22):2716-24. doi: 10.1001/archinte.163.22.2716. PMID 14662625
- [Background] Tulner LR, Frankfort SV, Gijsen GJ, van Campen JP, Koks CH, Beijnen JH. Drug-drug interactions in a geriatric outpatient cohort: prevalence and relevance. Drugs Aging. 2008;25(4):343-55. doi: 10.2165/00002512-200825040-00007. PMID 18361544
- [Background] Bates DW, Leape LL, Cullen DJ, Laird N, Petersen LA, Teich JM, Burdick E, Hickey M, Kleefield S, Shea B, Vander Vliet M, Seger DL. Effect of computerized physician order entry and a team intervention on prevention of serious medication errors. JAMA. 1998 Oct 21;280(15):1311-6. doi: 10.1001/jama.280.15.1311. PMID 9794308
- [Background] Durieux P, Trinquart L, Colombet I, Nies J, Walton R, Rajeswaran A, Rege Walther M, Harvey E, Burnand B. Computerized advice on drug dosage to improve prescribing practice. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD002894. doi: 10.1002/14651858.CD002894.pub2. PMID 18646085
- [Background] Egger T, Dormann H, Ahne G, Runge U, Neubert A, Criegee-Rieck M, Gassmann KG, Brune K. Identification of adverse drug reactions in geriatric inpatients using a computerised drug database. Drugs Aging. 2003;20(10):769-76. doi: 10.2165/00002512-200320100-00005. PMID 12875612
- [Background] Blix HS, Viktil KK, Moger TA, Reikvam A. Identification of drug interactions in hospitals--computerized screening vs. bedside recording. J Clin Pharm Ther. 2008 Apr;33(2):131-9. doi: 10.1111/j.1365-2710.2007.00893.x. PMID 18315778
- See also: Software to check multiple drug interactions. (Needs registration) — http://www.medscape.com/druginfo/druginterchecker
- See also: Free software in spanish to check drug interactions on line — http://www.medicamentosrothlin.com.ar/